CLINICAL TRIAL: NCT06661590
Title: Comparative Analysis Between Artificial Intelligence vs. Human Generated Nutrition Messages for Colorectal Cancer Survivors
Brief Title: Nutritional Language Model
Acronym: NLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00023189
Record Dates: First submitted 2024-10-15; First posted 2024-10-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: No Disease State or Condition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietician (Experimental)
  Interventions: Other: Nutritional Messaging

INTERVENTIONS:
Other: Nutritional Messaging — Dieticians will evaluate nutritional messages created by LLM and Human Experts.

SUMMARY:
Colorectal cancer survivors often face unique nutritional challenges and require support in their recovery and long0term health. While human experts have traditionally provided that support, there has been an increase in the use of Large Language Models (LLM) in medicine and in nutrition. The LLM offers a potential supplementary resource for generating personalized nutritional advice, specifically in personalized messaging. However, the efficacy and reliability of these AI-generated messages in comparison to human expert advice remain underexplored specific to this population.

This study aims to compare the nutrition-related content generated by popular LLMs-ChatGPT, Claude, Gemini, and Co-Pilot-against messages crafted by human experts. By evaluating the generated content in terms of readability, thematic relevance, medical relevance, perceived effectiveness, and implementation of participants' clinical practice, this research will provide insights into the strengths and limitations of using AI for nutritional guidance in colorectal cancer care.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Currently practicing Registered Dietitian Nutritionist with at least five years of experience working with oncology patients and survivors in their practice.
* Must have access to computer and internet access.

Exclusion Criteria:

* Non-English speakers, as the study materials and assessments are in English.
* Experts with conflicts of interest related to any of the LLMs that are being evaluated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Outcome Measure Title: Readability of Nutrition Messages | 8 to 12 months
  Description: The readability of AI-generated and human expert-generated nutrition messages will be measured using the Flesch-Kincaid Grade Level tool.
  Unit of Measure: Grade level score (numerical score indicating reading difficulty level).
  Measurement Tool: Flesch-Kincaid Grade Level formula. Scale values: The values vary from 0 to 18, where 18 represents the most difficult text.
Outcome Measure Title: Thematic Relevance of Nutrition Messages | 8 to 12 months
  Description: Thematic relevance of nutrition messages will be assessed by experts in nutrition using a thematic coding framework specifically designed for this study.
  Unit of Measure: Percentage (%) of messages that align with pre-determined thematic codes relevant to colorectal cancer survivorship.
  Measurement Tool: Thematic coding framework created by the research team. Scale values: The themes are capability (C), opportunity (O), and motivation (M) as three key factors capable of changing behavior (B).
Outcome Measure Title: Medical Relevance to Colorectal Cancer Survivors | 8-12 months
  Description: Medical relevance will be rated by specialists using a 0-5 relevance rating scale.
  Unit of Measure: Mean relevance score (0-5). Measurement Tool: Dietitians/Participants review using a relevance rating scale.
  Scale value: 1-5 (1- least, 5- most)
Outcome Measure Title: Perceived Effectiveness of Nutrition Messages | 8-12 months
  Description: Perceived effectiveness will be measured using a mean relevance score (1-5) administered to dietitians and participants.
  Unit of Measure: Mean relevance score (1-5). Measurement Tool: Dietitians/Participants survey. Scale value: 1-5 (1- least, 5- most)
Outcome Measure Title: Potential for Implementation in Clinical Practice | 8-12 months
  Description: Feasibility for clinical implementation will be rated by dietitians using a 1-5 feasibility scale.
  Unit of Measure: Mean feasibility score. Measurement Tool: Dietitians/Participants survey. Scale value: 1-5 (1- least, 5- most)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Lin, RD, PhD, Principal Investigator — Hormel Institute; Glen Morris, PhD, Study Chair — Hormel Institute
Locations (1):
- The Hormel Institute - University of Minnesota, Medical Research Center, Austin, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing the list of participation. This is due to the expected low enrollment amount of 6 participants.

REFERENCES:
- [Background] Shah NH, Entwistle D, Pfeffer MA. Creation and Adoption of Large Language Models in Medicine. JAMA. 2023 Sep 5;330(9):866-869. doi: 10.1001/jama.2023.14217. PMID 37548965
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37548965/